CLINICAL TRIAL: NCT00771524
Title: Open-Label, Pharmacokinetic Study of the Penetration of Ceftobiprole Into Bone
Brief Title: Pharmacokinetic Study of the Penetration of Ceftobiprole in the Bone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CR014227; PED-1001 (Other: Basilea Internal Reference)
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Total Hip Replacement Surgery
Keywords: Pharmacokinetics; Hip replacement; Ceftobiprole
MeSH Terms: interventions — ceftobiprole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceftobiprole (Experimental): Ceftobiprole, 500 mg single 2 hour infusion prior to hip replacement surgery
  Interventions: Drug: Ceftobiprole
- Control (No Intervention): Standard of care antibiotics prior to hip replacement surgery

INTERVENTIONS:
Drug: Ceftobiprole — Ceftobiprole, 500 mg single 2 hour infusion prior to hip replacement surgery
  Arms: Ceftobiprole

SUMMARY:
This study is being performed to measure the amount of the antibiotic ceftobiprole (study drug) found in the bone and blood after receiving one dose prior to your elective hip replacement surgery. A piece of your hip bone which will be removed as part of your surgery will be analyzed to determine how much ceftobiprole gets into the bone.

DETAILED DESCRIPTION:
About 20 patients will take part in the study. Two patients will not receive ceftobiprole, but will receive an antibiotic that is normally given prior to elective hip replacement surgery. The remaining 18 patients will receive ceftobiprole 500 mg dripped into the vein over 2 hours. All patients will have a sample of bone taken during the surgery and blood samples taken at specific timepoints. The samples taken from the 2 patients who did not receive study drug will assist in the development of a test used to measure the study drug in the bone sample. This is an open-label, parallel group, pharmacokinetic study in healthy men and women who have been cleared medically for elective total hip replacement surgery. Healthy is defined as patients who are medically stable and cleared for elective surgery. The study has 4 phases: a screening phase of up to 21 days before the day of surgery; a pretreatment phase of up to 7 days before the day of surgery; a 1-day open-label treatment phase; an end-of-study phase (end-of-study procedures or at the time of early withdrawal); and a follow-up telephone contact approximately 1 week after the surgery to assess new and ongoing adverse events. Two control subjects will be enrolled; these patients will not receive ceftobiprole, but will undergo surgery and a bone sample, which will serve as a control for qualifying the bioanalytical assay. The remaining 36 patients will be randomized to 1 of 2 ceftobiprole treatments. The primary objective is to estimate the penetration of ceftobiprole into bone of otherwise healthy patients who are undergoing total hip replacement surgery. Safety and tolerability will also be assessed. Venous blood samples will be collected and analyzed for ceftobiprole concentrations using validated liquid-chromatography methodology, with tandem mass spectrometric detection. Bone samples will be analyzed for ceftobiprole by qualified liquid-chromatography methodology, with tandem mass spectrometric detection. Safety and tolerability will be evaluated throughout the study. Blood will be drawn for clinical laboratory tests and PK evaluations. A single dose of ceftobiprole 500 mg dripped into the vein over 2 hours, administered prior to elective hip replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women at least 18 years of age who have elected to undergo hip replacement surgery. Subjects must be in overall good health with normal renal function (a creatinine clearance of >50 mL/min).

Exclusion Criteria:

* Subjects must not have a history of repeated severe nausea with anesthesia, gastric or duodenal ulcer, allergy to b lactam antibiotics, urinary obstruction or difficulty in voiding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The primary objective is to estimate the penetration of ceftobiprole into bone in otherwise healthy patients who are undergoing total hip replacement surgery. | 1 week

SECONDARY OUTCOMES:
Safety and tolerability will also be assessed. | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Ortho-McNeil Janssen Scientific Affairs, LLC